CLINICAL TRIAL: NCT05119686
Title: A Phase 2b, Randomized, Placebo-Controlled, Multicenter Study to Evaluate the Safety and Efficacy of AR882 Versus Placebo in Gout Patients
Brief Title: Phase 2b Evaluation of Efficacy and Safety of AR882 in Gout Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arthrosi Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AR882-202
Record Dates: First submitted 2021-10-20; First posted 2021-11-15 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Gout; Arthritis, Gouty; Hyperuricemia; Gout Chronic
MeSH Terms: conditions — Gout; Arthritis, Gouty; Hyperuricemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): AR882 Dose 1 x 12 weeks
  Interventions: Drug: AR882 Dose 1
- Group 2 (Experimental): AR882 Dose 1 x 2 weeks, then Dose 2 x 10 weeks
  Interventions: Drug: AR882 Dose 1; Drug: AR882 Dose 2
- Group 3 (Placebo Comparator): AR882 matching placebo x 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AR882 Dose 1 — Solid Oral Capsule
  Arms: Group 1; Group 2
Drug: AR882 Dose 2 — Solid Oral Capsule
  Arms: Group 2
Drug: Placebo — Matching Solid Oral Capsule Placebo
  Arms: Group 3

SUMMARY:
This study will assess the serum uric acid lowering effect and safety of AR882 in gout patients at two doses compared to placebo over 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* History of gout
* sUA > 7 mg/dL
* Estimated Glomerular Filtration Rate (eGFR) ≥ 30 mL/min/1.73m2

Exclusion Criteria:

* Malignancy within 5 years, except for successfully treated basal or squamous cell carcinoma of the skin
* History of cardiac abnormalities
* History of kidney stones

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2022-11-17 (Actual)

PRIMARY OUTCOMES:
Serum urate (uric acid) (sUA) level < 6 mg/dL following 6 weeks of dosing | 6 weeks
  Comparison of the treatment groups for the proportion of patients with serum urate (uric acid) (sUA) level < 6 mg/dL following 6 weeks of dosing

SECONDARY OUTCOMES:
sUA levels < 5, < 4, and < 3 mg/dL | 6 weeks
  Comparison of the treatment groups for proportion of patients whose sUA levels are < 5, < 4, and < 3 mg/dL
Incidence of Adverse Events | 14 weeks
  Treatment Emergent Adverse Events and Serious Adverse Event incidence.
Maximum Observed Plasma Concentration (Cmax) | 12 weeks
  Plasma samples will be collected to assess plasma concentrations at a series of timepoints to derive Cmax.
Time to observed Cmax (Tmax) | 12 weeks
  Plasma samples will be collected to assess plasma concentrations at a series of timepoints to derive Tmax.
Area under the plasma concentration-time curve (AUC) | 12 weeks
  Plasma samples will be collected to assess plasma concentrations at a series of timepoints to derive AUC.

CONTACTS AND LOCATIONS:
Overall Officials: R Keenan, MD, Study Chair — Arthrosi Therapeutics
Locations (22):
- United States (15):
  - Arthrosi Investigative Site, Gilbert, Arizona
  - Arthrosi Investigative Site, Sun City, Arizona
  - Arthrosi Investigative Site, Tucson, Arizona
  - Arthrosi Investigative Site, Miami, Florida
  - Arthrosi Investigative Site, Miami Lakes, Florida
  - Arthrosi Investigative Site, Tampa, Florida
  - Arthrosi Investigative Site, Honolulu, Hawaii
  - Arthrosi Investigative Site, Overland Park, Kansas
  - Arthrosi Investigative Site, Cleveland, Ohio
  - Arthrosi Investigative Site, Duncansville, Pennsylvania
  - Arthrosi Investigative Site, Dallas, Texas
  - Arthrosi Investigative Site, Houston, Texas
  - Arthrosi Investigative Site, Tomball, Texas
  - Arthrosi Investigative Site, West Jordan, Utah
  - Arthrosi Investigative Site, Glendale, Wisconsin
- Australia (2):
  - Arthrosi Investigative Site, Melbourne, Camberwell
  - Arthrosi investigative Site, Botany, New South Wales
- Taiwan (5):
  - Arthrosi Investigative Site, Taichung
  - Arthrosi Investigative Site - 301, Taipei
  - Arthrosi Investigative Site - 304, Taipei
  - Arthrosi Investigative Site, Taipei
  - Arthrosi Investigative Site, Taoyuan District